CLINICAL TRIAL: NCT05814484
Title: An Observational Cohort Study of Inhaler Adherence and Blood Eosinophil Count in Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Role of Inhaler Adherence and Blood Eosinophil Count in Exacerbations of COPD
Acronym: INCLINE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Leicester (Other)
Collaborators: Aparito Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 0884
Record Dates: First submitted 2023-03-22; First posted 2023-04-14 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Adherence, Treatment
Keywords: Blood Eosinophil Count; Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Full Blood Count (Plasma, Serum) Nasopharyngeal swab Urine Sputum C Reactive Protein
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study examining inhaler adherence and subsequent changes in blood eosinophil count in exacerbations of Chronic obstructive pulmonary disease (COPD) population.

The study will run for 6 months as an observation period. Passive inhaler adherence monitoring will be done electronically via inhaler sensors connected to mobile Apps, and collecting symptoms questionnaires, diary of exacerbation events and trial visits predominantly in remote fashion. It will explore the feasibility of digital platform in clinical practice to collect the adherence data along with exacerbation events.

DETAILED DESCRIPTION:
How Chronic Obstructive Pulmonary Disease (COPD) affects patients varies greatly among individuals. The concept of treatable traits, which identifies factors within an individual to allow targeted treatment has altered management strategies. The most commonly used biomarker for exacerbations of COPD is the blood eosinophil count [BEC], which tends to indicate a higher risk of exacerbations, but importantly is a biomarker of treatment response for corticosteroids.

Current pharmacological treatment for COPD is predominately based around inhaled therapy in the form of bronchodilators and inhaled corticosteroids (ICS) therapy.

However, almost half of the COPD population have been shown to poorly follow the prescribed inhaled therapy. This is important as a non-adherent trait may impact on BEC and result in unnecessary treatment escalation, increased risk to higher risk individuals (e.g. patients with high BEC) and lack of intervention around inhaler adherence.

Recent developments of digital platforms could potentially address this by capturing objective adherence data, unrecorded exacerbation events or if possible, anticipating the latter.

In summary, it is important to align inhaler adherence in conjunction with established biomarker, as is likely to help gain maximum benefit and better target interventions. In this study, the investigators propose the electronic monitoring of adherence and exacerbation reporting data along with the reflected changes in biomarkers and disease outcomes to lead a meaningful treatable trait approach in real-life setting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD documented by a health care provider with previous documented obstructive spirometry
* History of frequent exacerbations (defined as 2 or more exacerbations requiring oral corticosteroids and/or antibiotics within 12 months of pre-screening).
* Male or female participants aged ≥18 years.
* Willing and able to consent to participate in study.
* Able to use a smartphone device and comply with trial procedures.
* Participants with established triple therapy (ICS +LABA + LAMA) as controller at least 4 weeks prior to screening

Exclusion Criteria:

* Unable to give informed consent.
* Unable to use a smartphone device.
* Current or within the last 6 months (or maximum relevant wash out period, whichever is longer), participation in an investigational medicinal product (IMP) or device trial at the time of screening.
* Use of maintenance systemic corticosteroids within last 30 days.
* Patients whose treatment is considered palliative (life expectancy <6 months).
* History of unstable or severe cardiac, hepatic, or renal disease, or other medically significant illness, which the investigator believes, would be a contraindication to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with frequent exacerbation events
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Total number of exacerbation events | 24 weeks
  All exacerbation events during study period

SECONDARY OUTCOMES:
Number of participants who successfully completed the trial digital tasks | Month 6
  Participants who filled out electronic questionnaires and weekly symptom diaries
Feasibility of digital platform | Month 6
  Number of exacerbation events captured by digital platform
Change in blood eosinophil count over time | Month 1, 2,4 & 6
  Peripheral blood eosinophil count
Change in lung function test | Month 0 & 6
  Post-bronchodilator Forced Expiratory Volume in 1 second (FEV1)
Change in score of St George's Respiratory Questionnaire (SGRQ) | Month 0,2,4 & 6
  This 50-item questionnaire measures health status (quality of life) in patients with diseases of airway obstruction. Scores are broken down into 'symptoms' (normal participant range 9-15), 'activity' (normal participant range 7-12), 'impacts' (normal participant range 1-3), and a total score (normal participant range 5-7). Higher scores indicate poorer health status.
Change in score of COPD Assessment Tool (CAT) | Month 0,2,4 & 6
  The COPD Assessment Test (CAT) is a questionnaire for people with Chronic Obstructive Pulmonary Disease (COPD). It is designed to measure the impact of COPD on a person's life, and how this changes over time. Scores range from 0-40, with higher scores indicating greater impact of COPD on a patient's life.
Change in Extended MR dyspnoea score (eMRC) | Month 0,2,4 & 6
  This scale measures perceived respiratory disability. Participants rate their grades of breathlessness on a scale of 1 (least) to 5 (worst). The extension divides the grade 5 rating into 'a' (independent) and 'b' (dependent) to establish dependence on others for washing and dressing.
Number of exacerbation events | Month 6
  To compare between T2H and non T2H groups regardless of adherence level
Changes in blood eosinophil count | Month 1,2,4 & 6
  Comparison between nonT2high and T2high subgroups regardless of adherence rate

CONTACTS AND LOCATIONS:
Overall Officials: Neil Greening, Principal Investigator — University of Leicester, Biomedical Research Centre, Respiratory Science
Locations (1):
- NIHR Biomedical Research Centre, University of Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No